CLINICAL TRIAL: NCT06978244
Title: A Study to Assess Safety, Tolerability, and Pharmacokinetics of Ascending Concentrations of Topical Ocular BL1332 in Healthy Volunteers
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: BL-RX01-BL1332-1101
Record Dates: First submitted 2025-05-08; First posted 2025-05-18 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Ocular Pain
MeSH Terms: conditions — Eye Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BL1332 ophthalmic solution (0.06%, 0.15%, and 0.30% concentrations) (Experimental): BL1332 ophthalmic solution (0.06%, 0.15%, and 0.30% concentrations) administered as topical ocular drops
  Interventions: Drug: BL1332 ophthalmic solution
- BL1332 vehicle (Placebo Comparator): BL1332 vehicle administered as topical ocular drops
  Interventions: Drug: BL1332 ophthalmic vehicle

INTERVENTIONS:
Drug: BL1332 ophthalmic solution — Both arms taken four times a day for 1 day
  Arms: BL1332 ophthalmic solution (0.06%, 0.15%, and 0.30% concentrations)
Drug: BL1332 ophthalmic vehicle — Both arms taken four times a day for 1 day
  Arms: BL1332 vehicle

SUMMARY:
Single-Center, Phase 1 study to assess the ocular and systemic safety and tolerability of ascending concentrations of topical BL1332 ophthalmic solution eye drops compared with BL1332 vehicle in healthy volunteers, identifying the highest tolerated doses (HTDs)

DETAILED DESCRIPTION:
To assess the ocular and systemic safety and tolerability of ascending concentrations of topical BL1332 ophthalmic solution eye drops compared with BL1332 vehicle in healthy volunteers, identifying the highest tolerated doses (HTDs)

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent prior to conduct of any study-related assessment
2. Male and female subjects ≥18 to ≤50 years of age and in good health, as assessed by the Investigator from past medical history, physical examination, and laboratory tests at Screening
3. Vital signs assessed in the sitting position after the subject has rested for at least 3 minutes, within the following ranges at Screening and at the Baseline Visit:

   * Oral body temperature ≥35.0°C and ≤37.5°C
   * Systolic blood pressure ≥90 and <140 mmHg
   * Diastolic blood pressure ≥50 and <90 mmHg
   * Pulse rate ≥40 and ≤100 bpm
4. Body weight ≥50 kg
5. Body mass index (BMI) between 18.0 and 30.0 kg/m2 [BMI = Body weight (kg) / Height (m)2]
6. Corrected visual acuity of 20/40 (Snellen) or better in each eye at Screening
7. Able to communicate well with the Investigator and to understand and comply with the requirements of the study

Exclusion Criteria:

1. Women of childbearing potential (WOCBP) or non-vasectomized males with partners of childbearing potential are not eligible, unless they are using an effective method of contraception and agree to use an effective method of contraception until at least 30 days after study treatment.

   1. Women are considered of childbearing potential unless they have undergone permanent sterilization (such as hysterectomy, bilateral oophorectomy, bilateral salpingectomy, or bilateral tubal occlusion) or have been amenorrheic for ≥12 months without an alternative medical cause.
   2. Effective methods of contraception include systemic hormonal (inhibition of ovulation not primary mode of action) containing progestins only; single barrier male or female condom with or without spermicide or cap; diaphragm; sponge with spermicide; double barrier (male condom combined with one of the barrier methods); or intrauterine device
   3. Women who are pregnant, lactating, or breastfeeding are excluded.
2. Any medical condition (systemic or ophthalmic) that may, in the opinion of the Investigator and based on the content of the Investigator's Brochure (IB), preclude the safe administration of IP or safe participation in this study
3. Use of gabapentinoids or opioids within 30 days prior to Screening
4. Use of topical capsaicin within 30 days prior to Screening
5. Chronic use (defined as ≥15 days/month for 3 months prior to Screening) of acetaminophen or nonsteroidal anti-inflammatory drugs (NSAIDs) or anticipated regular (daily) use during the study
6. Chronic use of medications or dietary supplements (over-the-counter and/or prescription) that have not been stable for ≥14 days prior to Screening or any anticipated change in the chronic medication regimen
7. Reported use of tobacco products within 3 months prior to Screening and/or urine cotinine level consistent with use of tobacco product (not passive exposure) at Screening
8. History of use of marijuana/cannabinoid (CBD) or illicit substances including cocaine, heroin, methamphetamine, hallucinogens, or non-prescribed opioids within 3 months prior to Screening
9. Use of systemic corticosteroids, anticoagulants, or migraine medications such as ergotamine, calcitonin gene-related peptide (CGRP) antagonists within 30 days prior to the Baseline Visit
10. Use of cytochrome P450 3A4 (CYP3A4) or CYP3A5 inhibitors or inducers within 2 weeks prior to the Baseline Visit
11. History of any ocular surgery or ocular laser intervention within 6 months prior to Screening
12. History of any chronic eye disease other than refractive error, incipient cataract, strabismic amblyopia, or anisometropic amblyopia. Subjects with a history of acute eye disease (such as infection, corneal abrasion, or allergy) within 6 months prior to Screening may be eligible if the disease is not currently active.
13. Any currently active ocular condition that requires use of topical eye drops
14. Contact lens use within 2 weeks prior to Screening and throughout the study
15. Consumption of alcohol within 48 hours prior to the Baseline Visit and throughout the study
16. Donation or loss of ≥450 mL of blood within 8 weeks prior to Screening or longer, if required by local regulation
17. Hemoglobin <11.0 g/dL at Screening
18. Current or past history of human immunodeficiency virus (HIV) disease and/or hepatitis
19. Past participation in a clinical study within 30 days prior to Screening

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2025-07-29 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of DLTs (dose-limiting toxicities) | Approximately 6 months
  To assess the ocular and systemic safety and tolerability of ascending concentrations of topical BL1332 ophthalmic solution eye drops compared with BL1332 vehicle in healthy volunteers, identifying the highest tolerated doses (HTDs)
Incidence of treatment-emergent AEs (TEAEs) | Approximately 6 months
  To assess the ocular and systemic safety and tolerability of ascending concentrations of topical BL1332 ophthalmic solution eye drops compared with BL1332 vehicle in healthy volunteers, identifying the highest tolerated doses (HTDs)
Treatment-emergent changes in systemic and ocular safety assessments | Approximately 6 months
  To assess the ocular and systemic safety and tolerability of ascending concentrations of topical BL1332 ophthalmic solution eye drops compared with BL1332 vehicle in healthy volunteers, identifying the highest tolerated doses (HTDs)
PK profiles and following parameter, where data allow (Cmax) | Approximately 6 months
  To characterize the plasma PK after ocular administration of BL1332 in healthy volunteers
PK profiles and following parameter, where data allow ( Tmax) | Approximately 6 months
  To characterize the plasma PK after ocular administration of BL1332 in healthy volunteers
PK profiles and following parameter, where data allow (Ctau) | Approximately 6 months
  To characterize the plasma PK after ocular administration of BL1332 in healthy volunteers
PK profiles and following parameter, where data allow (Tlast) | Approximately 6 months
  To characterize the plasma PK after ocular administration of BL1332 in healthy volunteers
PK profiles and following parameter, where data allow ( AUClast) | Approximately 6 months
  To characterize the plasma PK after ocular administration of BL1332 in healthy volunteers
PK profiles and following parameter, where data allow (AUCtau) | Approximately 6 months
  To characterize the plasma PK after ocular administration of BL1332 in healthy volunteers
PK profiles and following parameter, where data allow (AUCinf) | Approximately 6 months
  To characterize the plasma PK after ocular administration of BL1332 in healthy volunteers
PK profiles and following parameter, where data allow (ke1) | Approximately 6 months
  To characterize the plasma PK after ocular administration of BL1332 in healthy volunteers
PK profiles and following parameter, where data allow (t1/2) | Approximately 6 months
  To characterize the plasma PK after ocular administration of BL1332 in healthy volunteers

CONTACTS AND LOCATIONS:
Locations (1):
- Site 101, Fair Lawn, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No